CLINICAL TRIAL: NCT02000661
Title: A Randomized Comparative Effectiveness Study of Routine Versus Selective Use of Fractional Flow Reserve (FFR) to Guide Non-Emergent Percutaneous Coronary Intervention (PCI)
Brief Title: Routine Versus Selective Use of FFR to Guide PCI
Acronym: FFR-SELECT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped early by DSMB due to slow enrollment - obtained data to be analyzed
Sponsor: Cardiology Research UBC (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Fung, MD, Principal Investigator, Cardiology Research UBC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H13-02709
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Acute Coronary Syndrome; Coronary Atherosclerosis; Angina, Unstable
Keywords: Fractional Flow Reserve (FFR); FFR guided coronary interventions; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine use of FFR (Experimental): Fractional Flow Reserve (FFR) used in most cases to guide PCI
  Interventions: Device: Fractional Flow Reserve (FFR)
- Selective use of FFR (Active Comparator): Fractional Flow Reserve (FFR) used at investigator discretion (Current practice)
  Interventions: Device: Fractional Flow Reserve (FFR)

INTERVENTIONS:
Device: Fractional Flow Reserve (FFR) — Fractional Flow Reserve (FFR) performed per guidelines to guide PCI
  Other Names: FFR Wire (PressureWire™ by St. Jude Medical)

SUMMARY:
Fractional flow reserve (FFR) is a test that can be performed at the time of heart catheterization. It measures the change in pressure across a narrowing in the heart artery during high flow situation, and provides reliable information about the functional severity of the narrowing. FFR measurements accurately predict whether a stent is needed, and is considered an excellent test before placement of stents to treat narrowed heart arteries. However, FFR is not used in every case because of the extra time needed and the associated device costs. Cardiac Services BC (an agency of Provincial Health Services Authority) is sponsoring this study to find out if FFR should be used in most cases (routine), rather than the current selective approach.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is an effective, less invasive mode of revascularization compared with coronary artery bypass grafting (CABG). In 2011, a total of 7,614 PCI procedures were performed in British Columbia (BC). While some procedures were done emergently for life-threatening indications (e.g. ST elevation myocardial infarction - STEMI or cardiogenic shock), most (6,169 cases in year 2011) were done at the discretion of the treating physicians, taking patient preference into account. A number of factors are usually considered before proceeding with PCI. These may include clinical presentation (stable angina versus acute coronary syndrome); severity of symptoms (asymptomatic or highly symptomatic); response to medical therapy; severity of ischemia based on non-invasive functional testing (mild, moderate, or severe); predicted risk (low, intermediate, or high); and findings on coronary angiography (lesion number, location, severity, and morphology, etc). However, interpretation of symptoms is subjective. Non-invasive tests for ischemia may not be reliable. In addition, coronary angiography uses 2 dimensional images to depict 3-dimensional structures, and there is well known limitations.

The concept of using fractional flow reserve (FFR) to predict the functional significance of coronary lesions was described > 20 years ago. In 1996, Pijls et al showed that measurements of FFR in the cardiac catheterization laboratory can accurately predict provoked ischemia upon non-invasive functional testing. The DEFER study (2007) showed that coronary lesions with non-ischemic FFR values can be treated with medical therapy with good clinical outcome at 5-year follow up. The FAME-1 study (2009) evaluated the strategy of PCI guided by angiography versus PCI guided by FFR measurements in multi-vessel disease. The primary end-point was the 1-year composite of death, myocardial infarction (MI), and any repeat revascularization. Fewer stents were used per patient for the FFR-guided group (2.7 versus 1.9 stents per patient), less contrast agent used (302 versus 272 ml), and lower in-lab equipment cost ($6,007 US versus $5,332 US), all significant with P<0.001. A total of 1,005 patients were randomized. At 1-year follow up, the composite end-point of death, MI and target vessel revascularization was 18.2% for the angiography-guided group versus 13.3% for the FFR-guided group (p < 0.02). At 2-year follow up, the incidence of death and MI was lower for the FFR-guided group (12.7% versus 8.4%, p<0.03), and the incidence of MI in the FFR-guided and PCI deferred population was very low at 0.2%.

Since the publication of the FAME-1 study, the use of pressure wires to measure FFR increased from ~400 cases per year to ~1,000 cases per year in BC. However, in comparison with an annual non-emergent PCI volume of >6,000 cases per year, the use of FFR appears highly selective (1,058 out of 6,169, 17%, based on year 2011 statistics). In a series of 442 consecutive FFR cases done at the Vancouver General and St. Paul's Hospitals (year 2011 to 2012), the use of FFR identified non-ischemic lesions in 52%, and this resulted in a change in management decision in 68%. In addition, provincial data showed significant variation in the use of FFR among the 5 PCI capable hospitals in BC (from <5% to ~30%). Based on the recent European Society of Cardiology guidelines, the use of FFR to guide revascularization has a class 1a indication in multi-vessel disease, while the US guidelines (American College of Cardiology, ACC) has a class 2a recommendation for the use of FFR in evaluating coronary lesions of intermediate severity. It is possible that a highly selective approach to the use of FFR may lead to underuse, which in turn may lead to overuse of PCI, with increased cost, and adverse clinical outcome.

We hypothesize that the routine use of FFR may improve clinical outcome, decrease the number of PCI, and decrease direct cost in the cardiac catheterization laboratory. We propose a randomized study to compare 2 approaches of using FFR to guide PCI: (1) routine use - the experimental arm; and (2) selective use - the current standard.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with stable coronary artery disease or recent acute coronary syndrome (ACS). Subjects who present with ST elevation myocardial infarction (STEMI) are allowed to be included after 5 days from initial presentation.
2. At least one obstructive coronary lesion is present with vessel reference diameter ≥2.5 mm and diameter stenosis ≥50% by visual estimate. Lesions must be technically suitable for the FFR procedure and angioplasty with stent placement.
3. Physician will classify all target lesions and need for FFR before randomization, and there is a plan to perform a non-emergent PCI.
4. Subject is ≥18 years old, with signed informed consent.

Exclusion Criteria:

1. Expected non-cardiac longevity < 2 years.
2. Planned treatment with CABG.
3. Planned treatment with medical therapy.
4. Left main disease > 50% diameter stenosis based on visual estimate.
5. Safety issues:

   1. Unstable hemodynamics or serious arrhythmias during procedure;
   2. Ongoing ischemic chest pain;
   3. High grade AV block (unless pacemaker);
   4. Allergic to adenosine.
6. When FFR is clearly not needed:

   1. Target vessel with slow flow (< TIMI-3);
   2. Single vessel disease with ≥90% stenosis;
   3. Single vessel disease with ≥80% stenosis and documented ischemia on functional imaging test;
   4. In acute coronary syndrome, ≥70 stenosis identified as culprit.
7. When FFR is clearly needed for all target lesions: as declared by the operator.
8. Technical difficulty:

   1. Severe vessel tortuosity;
   2. Severe coronary calcification;
   3. Anticipate difficult wiring;
   4. Aorto-ostial lesion (ok for IV adenosine is used as the hyperemic agent).
9. Interpretation difficulty:

   1. Target vessel acting as a major collateral donor;
   2. When RA pressure very high;
   3. STEMI within past 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2014-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Composite of all cause mortality, repeat hospitalization for MI or repeat revascularization (PCI or coronary artery bypass grafting - CABG) | 1 Year

SECONDARY OUTCOMES:
All cause mortality | 1 Year
Repeat hospitalization for MI | 1 Year
Rate of repeat revascularization (PCI or CABG) | 1 Year
Time of procedure, contrast amount, and radiation dose | Post-procedure

OTHER OUTCOMES:
Economic evaluation, including health resource utilization | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fung, MBBS, FRCPC, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - Kelowna General Hospital, Kelowna, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia